CLINICAL TRIAL: NCT05779553
Title: Evaluation of Serum Tumor Endothelial Marker 1 as a Potential Biomarker for Colorectal Cancer Diagnosis and Cancer Progression
Brief Title: Evaluation of Serum Tumor Endothelial Marker1 as a Potential Biomarker for Colorectal Cancer Diagnosis and Cancer Progression
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Esraa Emad Abdel Azeem Kamel, Assiut lecturer, Assiut University
Other Study IDs: HIJHN
Record Dates: First submitted 2023-01-14; First posted 2023-03-22 (Actual); Last update posted 2023-03-22 (Actual); Status verified 2023-03

CONDITIONS: Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group (1)(patient group):: who are 50 newly diagnosed patient with colorectal cancer, who will be admitted at South Egypt Cancer Inistitute and Assiut University Hospital during 2023.
  Patients group will be furtherly subclassified according to the American Joint Committee on Cancer Staging,TNM staging classification
  Interventions: Diagnostic Test: Tumor Endothelial Marker 1 ( TEM1 ) by ELISA kits
- Group (2) (control group): 40 apparently healthy individuals with matched age and sex are included in this study as a control group for comparison.
  Interventions: Diagnostic Test: Tumor Endothelial Marker 1 ( TEM1 ) by ELISA kits

INTERVENTIONS:
Diagnostic Test: Tumor Endothelial Marker 1 ( TEM1 ) by ELISA kits — measurement of serum TEM1 in CRC patients, its relation to staging and comparing the diagnostic performance of serum TEM1 with serum CEA and CA19-9 for diagnosis of CRC. and Early detection of CRC patient

SUMMARY:
Aim of work

1. measurement level of serumTEM1 in CRC patients by ng/ml using ELISA kits .
2. find relation between serum TEM1 level and staging of CRC patients .
3. measurement of serum CEA , CA19-9 levels by ng/ml so we can can compare their levels with serum TEM1 level in CRC patients .

DETAILED DESCRIPTION:
Colorectal cancer (CRC) is a serious health problem, a challenge for research, and a model for studying the molecular mechanisms involved in its development. Colorectal cancer is the third most common cancer in the world with approximately 1.4 million new cases and almost 700,000 associated deaths reported per year. The incidence, morbidity, and mortality rates of CRC are expected to increase due to population aging and profound adverse effects of many life style-related factors.

Tumor growth is dependent on the complex and multistage angiogenesis. Tumor blood vessels are characterized with abnormal morphology and function compared to normal blood vessels. Except for disorganized structure, abnormal basement membrane, and increased leakiness, tumor vascular cells express unique protein named (Tumor endothelial marker 1 (TEM1)- endothialin-CD248) .

Tumor endothelial marker is a transmembrane glycoprotein which expression is significantly higher in tumor vasculature (5-,10-, and 20-fold) compared to the vessels of healthy tissues. It was suggested TEMs could discriminate between tumor and nontumor vascular cells.

Tissue overexpression of TEM1 was found in patients with CRC compared to healthy controls as well as in rectal cancer tissues when comparing tumor, lymph nodes, metastasis (TNM) stage I with other stages: TNM II, III, IV , Although the biology of TEM1 is intensely studied, including clinical studies with anti-TEM1 molecules, Only one study (2020) determined the potential usefulness of serum TEM1 in CRC. Pietrzyk (2020) revealed that TEM1 demonstrated higher levels in the serum of the patients with CRC than healthy individuals and reported that TEM1 could act as a potential diagnostic, progression, and prognostic serum biomarker for patients with CRC. Most commonly used serum markers for diagnosis and monitoring of CRC are carcinoembryonic antigen (CEA) and carbohydrate antigen 19-9 (Ca 19-9). However, these markers show insufficient sensitivity, especially at early stages of CRC. Therefore, finding sensitive and specific, noninvasive, serum biomarkers is a prerequisite for early CRC diagnosis.

ELIGIBILITY:
Inclusion Criteria:

1-newly diagnosed CRC patients.

Exclusion Criteria:

1. chemotherapy
2. radiotherapy
3. surgical treatment
4. heart failure
5. angina
6. liver cirrhosis
7. renal cell carcinoma
8. gastric cancer.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: * Fifty patients who were diagnosed by (lower endoscopy, multislice CT abdomen or histopathology analysis of the lesion), tumor staging was classified according to the American Joint Committee on Cancer Staging,TNM staging classification.
  * Patients did not receive any chemotherapy or undergo surgical treatment
  * Forty apparently healthy individuals with matched age and sex are included in this study as a control group for comparison
Sampling Method: Non-Probability Sample
Enrollment: 90 (Estimated)
Dates: Start 2023-05-01 (Estimated); Primary Completion 2026-02-01 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Tumor endothelial marker 1 in colorectal cancer | baseline
  1. measurement level of serumTEM1 in CRC patients by ng/ml using ELISA kits .
  2. measurement of serum CEA , CA19-9 levels by ng/ml